CLINICAL TRIAL: NCT03866226
Title: The Effect of Ambulatory Blood Pressure Monitoring on Sleep Disturbance
Brief Title: The Effect of ABPM on Sleep Disturbance
Acronym: EMBED
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, XiaoHong PAN, PI, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: I2017001235
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Blood Pressure Monitoring, Ambulatory
Keywords: ambulatory blood pressure monitoring; sleep

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ambulatory blood pressure monitoring (ABPM) is an ideal tool for the diagnosis and evaluation of hypertension.However, ABPM frequently measures the tightening feeling and buzzing sound of the blood pressure cuff during nighttime, which can cause the patient to wake up easily during sleep, which will affect the sleep of the patient. Moreover, improper awakening of the patient from sleep can significantly increase the patient's blood pressure and affect the accuracy of ABPM monitoring. The Effect of ABPM on Sleep Disturbance (EMBED) study is designed to examine whether ABPM affects sleep, as well as the relationship and influencing factors of sleep and ABPM results, and screening for people who are susceptible to ABPM testing.

DETAILED DESCRIPTION:
Participants who accept ABPM in the Second Affiliated Hospital of Zhejiang University School of Medicine, will be recruited for EMBED enrollment. Participants will be asked to provide basic background information and to fill out the STOP-BANG evaluation form. Anxiety, depression, insomnia, sleep questionnaire and pain assessment scale for cuff inflation are used to assess characteristics of participants and their sleep quality. Before ABPM starts, office blood pressure of participants will be measured. Participants will undergo ABPM under standardized guidance. At the end of ABPM, participants will be asked to fill in sleep questionnaire and pain assessment scale for cuff inflation again. EMBED proposes to study whether ABPM affects sleep, as well as the relationship and influencing factors of sleep and ABPM results, and screening for people who are susceptible to ABPM testing. A better understanding of interaction between ABPM and sleep will help us further evaluate the accuracy of ABPM and more precisely control diurnal hypertension in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Age 18-80 years
3. Capable of understanding the test and cooperating with the questionnaire.

Exclusion Criteria:

1. History of psychosis, including schizophrenia, bipolar disorder, depression, anxiety, obsessive-compulsive disorder, phobia, somatoform disorder, stress-related disorders
2. History of insomnia, currently with medication
3. History of obstructive sleep apnea (OSA)
4. History of other sleep disorders, including narcolepsy/hypersomnias, circadian rhythm sleep disorder, parasomnias, sleep-related dyskinesia
5. History of heart failure, that is New York heart association (NYHA) Class Ⅲ-Ⅳ
6. History of atrial fibrillation and frequent atrial or ventricular extrasystoles
7. Ongoing substance or alcohol abuse
8. Currently receiving sedative hypnotic medication within 1 week
9. Pregnant women
10. Ongoing involvement in night-shift work (22:00-6:00) within 1 week
11. Ongoing need of care of families at home that wake during the night within 1 week
12. Incomprehensible or unwilling to fill in informed consent or questionnaire

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who undergo ABPM in the Second Affiliated Hospital of Zhejiang University School of Medicine
Sampling Method: Probability Sample
Enrollment: 564 (Actual)
Dates: Start 2019-03-10 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Sleep questionnaire score will be used to evaluate the alteration of sleep | about 2 days
  Sleep questionnaire score

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Qian N, Yang D, Li H, Ding S, Yu X, Fan Q, Yu Z, Ye S, Yu H, Wang Y, Pan X. Considering Psychosocial Factors When Investigating Blood Pressure in Patients with Short Sleep Duration: A Propensity Score Matched Analysis. Int J Hypertens. 2021 Nov 30;2021:7028942. doi: 10.1155/2021/7028942. eCollection 2021. PMID 34888099

DOCUMENTS (1):
  • Study Protocol (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT03866226/Prot_000.pdf